CLINICAL TRIAL: NCT01268982
Title: Dimensional Changes of the Alveolar Ridge Contour After Socket Preservation, Stability of Implants Placed, and Histological Evaluation of Newly Formed Bone at These Sites.
Brief Title: Effect of Socket Preservation Procedure on Dimensional Changes of the Ridge, and Its Efficacy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Dr. Hamidreza Arab, Mashhad Dental School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 88724
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-01

CONDITIONS: Alveolar Bone Atrophy
Keywords: socket preservation; alveolar ridge augmentation
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- preserved socket (Experimental): sockets will be filled with DFDBA and covered with absorbable membrane. Primary coverage will be achieved by full thickness mucosal flap advancement over each socket.
  Interventions: Procedure: socket preservation

INTERVENTIONS:
Procedure: socket preservation — sockets will be filled with DFDBA and covered with absorbable membrane. Primary coverage will be achieved by full thickness mucosal flap advancement over each socket
  Other Names: DFDBA

SUMMARY:
In this study, the investigators will evaluate the dimensional changes of alveolar bone in the preserved sites in comparison with extraction only conventional healed sockets, as well.

1. Dimensional changes of the alveolar ridge contour after socket preservation in comparison to conventional tooth extraction.
2. Evaluation the stability of implants placed at the preserved sockets.
3. Histological evaluation of newly formed bone at the socket preserved sites in comparison with extracted only healed sites.

DETAILED DESCRIPTION:
Nineteen systematically healthy patients (10 female and 9 male; mean age 38 years old; range 19-57) providing 32 hopeless non-molar teeth were selected and divided into 2 treatment groups: In the test group, following tooth extraction, for 16 sockets (9sockets from 5 female and 7 sockets from 5 male patients) soft and hard tissue measurements include horizontal (Bucco-Lingual dimensions at 1mm,3mm and 7mm at the mid portion from the line connecting two adjacent CEJs) and vertical ridge dimensions (vertical distance from the line connecting two adjacent CEJs at 8 points: Mid-Buccal, Mid-Lingual, Mesial, Distal, Disto-Buccal, Disto-Lingual, Mesio-Buccal, Mesio-Lingual around the socket) will be determined using a caliper and a template. All sockets will be filled with DFDBA and covered with absorbable membrane. Primary coverage will be achieved by full thickness mucosal flap advancement over each socket. Then an acid-etch bridge will be applied for the sites, both to avoid the movement of adjacent teeth to the empty space & also for patients esthetics. 6 months following the procedure, the soft and hard tissue in all the sites will be measured again as it was mentioned previously, plus the measurements gained from CBCT radiographs.

Besides, biopsy will be harvested from some of the preserved sites that has enough width with the use of trephine bur no.3 and it was sent for histological evaluation. Subsequently, Implants will be installed in the preserved sites and the implant stability will be measured with the help of Ostell device. The stability will be measured after 4 month following implant insertion with the same device while the implant undergoes the implant exposure procedure.

In control group, 16 sockets (9 sockets from 5 female, and 7 sockets from 4 male patients) served as unfilled extraction only group. Following extraction, soft and hard tissue measurements (horizontal and vertical ridge dimensions) will be determined with the use of caliper and template.

6month after extraction, CBCT will be taken from the site and at the time of implant installation, the soft and hard tissue in all sites will be measured in vertical and horizontal dimensions. Furthermore, biopsy from some of the healed sockets with enough width will be taken with the use of trephine bur no.3 and it will be sent for histological examination.

ELIGIBILITY:
Inclusion Criteria:

* Non-molar hopeless teeth
* lack of bone volume for ideal implant placement

Exclusion Criteria:

* Patient's un-wiliness for involvement in the project
* contraindication of surgery due to medically-related problems

Ages: 19 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
soft and hard tissue vertical and horizontal changes | 6 months
  soft and hard tissue measurements include horizontal (Bucco-Lingual dimensions at 1mm,3mm and 7mm at the mid portion from the line connecting two adjacent CEJs) and vertical ridge dimensions (vertical distance from the line connecting two adjacent CEJs at 8 points: Mid-Buccal, Mid-Lingual, Mesial, Distal, Disto-Buccal, Disto-Lingual, Mesio-Buccal, Mesio-Lingual around the socket)

SECONDARY OUTCOMES:
histologic evaluation and implant stability measurement | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: hamid reza arab, DDS.,Ms., Principal Investigator — Mashhad University of Medical Sciences
Locations (1):
- Mashhad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran